CLINICAL TRIAL: NCT02783612
Title: Improvement of Compliance by Digital Blood Glucose Monitoring of Women With Gestational Diabetes
Brief Title: Digital Glucose Monitoring in Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: GDMAPP
Record Dates: First submitted 2016-04-12; First posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glucose application (Experimental): Regular high risk pregnancy clinic surveillance in addition to a Smart phone application for registering the Blood glucose levels and submitting via email every 3-5 days to the High risk Doctor involved in the trial.
  Interventions: Other: glucose buddy application
- Regular monitoring (No Intervention): Regular high risk pregnancy clinic surveillance

INTERVENTIONS:
Other: glucose buddy application
  Arms: glucose application

SUMMARY:
Assessing blood glucose control in women with gestational diabetes can be challenging. The standard of care remains visual inspection of blood glucose paper diaries of self-performed capillary monitoring during regular meeting in High Risk pregnancy clinics.

The researchers are interested in preforming a randomized control trial comparing women with the diagnosis of gestational diabetes with regular High-Risk clinic surveillance to digital monitoring using an application in a Smart-phone and submitting those values via email in addition to the regular clinic appointments.

The Primary outcome of the trial is to assess the compliance of the research group as compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* gestational diabetes

Exclusion Criteria:

* pre-gestational diabetes

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Assessing the compliance of the research group compared to the control group. | 18 month
  By calculating the amount of daily glucose measurements in the research group compared to the number of glucose measurements in the control group

CONTACTS AND LOCATIONS:
Locations (1):
- Wolfson medical center, Holon, Israel

IPD SHARING:
Plan to Share IPD: Undecided